CLINICAL TRIAL: NCT03173599
Title: A Safety and Tolerability Evaluation of Ascending Single Oral Doses of Metacavir Enteric-coated Capsules Using a Randomized，Double-blind, Placebo-controlled Design Conducted in Chinese Healthy Adult Volunteers
Brief Title: The Safety and Tolerability of Metacavir Enteric-coated Capsules in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNA20100714
Record Dates: First submitted 2017-05-12; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Peptide Nucleic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- PNA 40mg (Experimental): Metacavir Enteric-coated Capsules,oral before meal
  The beginning dose is 40mg,If no adverse effects were observed in 40 mg, the next dose group was started of 80mg.
  Interventions: Drug: PNA 40mg
- PNA 80mg (Experimental): Metacavir Enteric-coated Capsules,oral before meal
  The single dose is 80mg,If no adverse effects were observed in 80 mg, the next dose group was started of 160mg.
  Interventions: Drug: PNA 80mg
- PNA 160mg (Experimental): Metacavir Enteric-coated Capsules,oral before meal
  The single dose is 160mg,If no adverse effects were observed in 160 mg, the next dose group was started of 240mg.
  Interventions: Drug: PNA 160mg
- PNA 240mg (Experimental): Metacavir Enteric-coated Capsules,oral before meal
  The single dose is 240mg,If no adverse effects were observed in 240 mg, the next dose group was started of 360mg.
  Interventions: Drug: PNA 240mg
- PNA 360mg (Experimental): Metacavir Enteric-coated Capsules,oral before meal
  The single dose is 360mg,If no adverse effects were observed in 360 mg, the next dose group was started of 480mg.
  Interventions: Drug: PNA 360mg
- PNA 480mg (Experimental): Metacavir Enteric-coated Capsules,oral before meal
  The single dose is 480mg.
  Interventions: Drug: PNA 480mg
- PNA Placebo (Placebo Comparator): Metacavir Enteric-coated Capsules Placebo,oral before meal
  The beginning dose is 40mg/d, the dose escalation method is 40mg/80mg/160mg/240mg/360mg/480mg
  Interventions: Drug: PNA Placebo

INTERVENTIONS:
Drug: PNA 40mg — The beginning dose is 40mg.
  Other Names: Metacavir Enteric-coated Capsules 40mg
  Arms: PNA 40mg
Drug: PNA 80mg — The single dose is 80mg.
  Other Names: Metacavir Enteric-coated Capsules 80mg
  Arms: PNA 80mg
Drug: PNA 160mg — The single dose is 160mg.
  Other Names: Metacavir Enteric-coated Capsules 160mg
  Arms: PNA 160mg
Drug: PNA 240mg — The single dose is 240mg.
  Other Names: Metacavir Enteric-coated Capsules 240mg
  Arms: PNA 240mg
Drug: PNA 360mg — The single dose is 360mg.
  Other Names: Metacavir Enteric-coated Capsules 360mg
  Arms: PNA 360mg
Drug: PNA 480mg — The single dose is 480mg.
  Other Names: Metacavir Enteric-coated Capsules 480mg
  Arms: PNA 480mg
Drug: PNA Placebo — The beginning dose is 40mg/d, the dose escalation method is 40mg/80mg/160mg/240mg/360mg/480mg.
  Other Names: Metacavir Enteric-coated Capsules Placebo
  Arms: PNA Placebo

SUMMARY:
A Safety and Tolerability Evaluation of Ascending Single Oral Doses of Metacavir Enteric-coated Capsules Using a Randomized，Double-blind, Placebo-controlled Design conducted in Chinese Healthy Adult Volunteers.

DETAILED DESCRIPTION:
A study to evaluate the safety and tolerability of ascending single oral doses of metacavir enteric-coated capsules using a placebo-controlled design conducted in Chinese healthy adult volunteers, and to provide references for the clinical trial of the next phase Ⅰ and Ⅱ.

48 eligible healthy subjects are involved. According to the set ascending-doses groups, subjects will be randomized in a 3:1 proportion to orally take a single dose of Metacavir enteric-coated capsule or placebo on the condition of fasting. Each group has 8 people, evenly composed of men and women. The beginning dose of the study is 40mg/d.According to the dose escalation method, subjects who have successfully completed tests of the previous dose group and passed the safety assessment will enter the next dose group with the same method. All subjects check in the phaseⅠresearch center one day early before taking the test drug. Vital signs and ECG will be observed before and 0.5,1,2,4,8,12,18,24,48,72 hours after administration and at the follow-up day which is the 7th day since administration. Laboratory tests will be conducted before and 6,24,48,72 hours after administration and at the follow-up day , and the adverse drug events are observed throughout the test.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 18 to 45 years old ;
2. Body mass index (BMI) above/equal 18 and below 28 kg/m2;
3. Child bearing potential, has a negative serum pregnancy test at screening period, and agrees to use contraceptions consistently and correctly in 14 days after dosing;
4. No smoking in a year before post-dosing of study drug;
5. Give their signed written informed consent to participate.

Exclusion Criteria:

1. Subjects who have clinically significant abnormal laboratory test results;
2. Subjects with clinically significant abnormal ECG;
3. Subjects with cardiac or blood disease affecting the safety and pharmacokinetics;
4. Subjects with liver or renal disease affecting the safety and pharmacokinetics;
5. Subjects with digestive system disease affecting the safety of study drug;
6. Subjects with other acute or chronic disease affecting pharmacokinetics and product metabolism;
7. A positive hepatitis B surface antigen, hepatitis C or HIV test result;
8. History of hypersensitivity or allergy to any of the study drugs or to drugs of similar chemical classes;
9. Subjects, who in the opinion of the investigator, significantly abuse alcohol;
10. Drink in 36 hours before post-dosing of study drug;
11. Ingest any foods or beverages which may affect pharmacokinetics;
12. Drug abuse,a history of poisoning;
13. Smokers(use tobacco products in a year before post-dosing of study drug);
14. Subjects who had received other medications within 2 weeks prior to the first administration of Investigational Product,and the original and main metabolites were not completely eliminated;
15. Subjects who participated in any other clinical trials within 3 months prior to the administration of Investigational Product;
16. Subjects who had suffered from hemorrhage or blood donation over 200ml will be excluded; 17. Subjects over exercised accompanied with fatigue and muscle aches within 1 week period to the administration of Investigational Product;

18．Children,women who are pregnant,lactating,with childbearing potential and who are using acyeterions; 19．Haven't given their signed written informed consent to participate; 20．Subjects in the opinion of the investigator, could not participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline, up to Day 7
  Adverse Events refer to any adverse and unexpected vital signs and laboratory tests，symptoms or temporary illness.

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Mao, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No